CLINICAL TRIAL: NCT00547092
Title: A Multicenter Open-Label Study to Determine Treatment Preference of Tadalafil (IC351, LY450190) or Sildenafil Citrate in the Oral Treatment of Erectile Dysfunction
Brief Title: Study For Which Treatment, Tadalafil or Sildenafil, is Preferred For Problems Getting or Maintaining an Erection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7002; H6D-MC-LVFL
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): tadalafil given the first 12 weeks and after a 4 week washout sildenafil is given for 12 weeks.
  Interventions: Drug: tadalafil
- 2 (Active Comparator): sildenafil given the first 12 weeks and after a 4 week washout tadalafil is given for 12 weeks.
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: tadalafil — 10 mg or 20 mg tadalafil tablets, as needed, no more than once a day, by mouth for 12 weeks (8 week treatment experience phase and a 4 week treatment assessment phase)
  Other Names: LY450190; Cialis; IC351
  Arms: 1
Drug: sildenafil — 25 mg, 50 mg, or 100 mg sildenafil citrate tablets, as needed, no more than once a day, by mouth for 12 weeks (8 week treatment experience phase and a 4 week treatment assessment phase)
  Arms: 2

SUMMARY:
To determine if men prefer tadalafil or sildenafil for getting and keeping an erection after treatment with both drugs.

ELIGIBILITY:
Inclusion Criteria:

* History of erection problems
* Never taken treatments known as PDE5 inhibitors for erection issues
* Abstain from using any other erection treatments during the study
* Anticipate a monogamous female sexual relationship
* Must be able to make required sexual intercourse attempts

Exclusion Criteria:

* History of other primary sexual disorder
* Treatment with nitrates
* Have a penile implant or clinically significant penile deformity
* History of certain heart problems
* Do not meet certain lab value reference ranges

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2003-10; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Preference Assessment measured by the Treatment Preference Question | 26 weeks

SECONDARY OUTCOMES:
Compare efficacies of the two drugs as measured by the Erectile Function domain of IIEF and Questions 2 and 3 of the SEP diary. | 0, 12, and 26 weeks
Assess sexual encounters attributes measured by the PAIRS. | 0, 12, and 26 weeks
Measure adverse events through the Side Effect Question. | 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, United Kingdom

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com